CLINICAL TRIAL: NCT03726398
Title: CompRehensive Phenotypic Characterization of Patients With Scleroderma-Associated Interstitial Lung DiseasE and Pulmonary Hypertension (PH): The CRuSADE PH Study
Brief Title: CompRehensive Phenotypic Characterization of Patients With Scleroderma-Associated ILD and PH
Acronym: CRUSADE
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Did not identify eligible candidates
Sponsor: Franz Rischard, DO (Other)
Collaborators: National Jewish Health (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Franz Rischard, DO, Associate Professor, Medicine, University of Arizona
Organization: University of Arizona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IIS-02801
Record Dates: First submitted 2018-10-21; First posted 2018-10-31 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Interstitial Lung Disease; Scleroderma; Pulmonary Hypertension
MeSH Terms: conditions — Lung Diseases, Interstitial; Scleroderma, Diffuse; Hypertension, Pulmonary | interventions — macitentan; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Opsumit (Experimental): Opsumit 10 mg tablet by mouth once daily
  Interventions: Drug: Opsumit 10 Mg Tablet

INTERVENTIONS:
Drug: Opsumit 10 Mg Tablet — Oral tablet taken once daily
  Other Names: Macitentan

SUMMARY:
Patients with interstitial lung disease (ILD) and scleroderma who develop pulmonary hypertension (PH) do not fit well into the current classification system and treatments for pulmonary hypertension. This study aims to better understand patients with ILD-PH and scleroderma and to determine if treatment with Macitentan is beneficial.

DETAILED DESCRIPTION:
The investigators aim to use pressure-volume loop derived right ventriculo-vascular coupling, pulmonary impedance, and invasive cardiopulmonary exercise testing (CPET) to:

1. Comprehensively phenotype patients with scleroderma ILD-PH and pulmonary vascular exercise limitation (PVL) relative to scleroderma ILD-PH without PVL.
2. Compare the efficacy of chronic Macitentan therapy in improving 1) right ventricular hemodynamics 2) exercise capacity and 3) symptoms in scleroderma ILD-PH patients with and without PVL.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have scleroderma ILD will be defined as having a total lung capacity of less than 80% predicted and CT evidence of fibrosis. The degree of fibrosis will be scored by a radiologist using the CT comparative scoring method of Wells et al (13).
* Pulmonary Hypertension (PH) as defined as resting mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg with a wedge pressure of ≤ 15 mmHg during right heart catheterization.
* Stable ILD as evident by a stable FEV1 and FVC for 3 months prior to the initiation of the study, and be pulmonary arterial hypertension (PAH)-targeted treatment naïve.

Exclusion Criteria:

* Patients with a left ventricular ejection fraction <50% or clinical, echocardiographic, and/or catheterization data consistent with heart failure with preserved ejection fraction (HFpEF) and/or moderate-severe aortic or mitral valve abnormality
* Patients with severe restrictive lung disease (FVC<40% predicted) and/or obstructive lung disease (FEV1 <55% predicted and FEV1/FVC <70%).
* Patients with radiographic combined pulmonary fibrosis/emphysema (CPFE) will also be excluded if imaging shows predominant emphysema and/or obstruction is moderately severe (FEV1<30%)
* Patients with a history of pulmonary embolism within the last three months or evidence of chronic pulmonary embolism.
* Patients with a known contraindication to right heart catheterization.
* Patients whom have received active or previous pulmonary vasoactive medication within the previous 12 weeks.
* Patients with a contraindication to exercise testing based on American Heart Association/American College of Cardiology (AHA/ACC) guidelines.
* PAH associated with significant venous or capillary involvement (PCWP > 15 mmHg), known pulmonary veno-occlusive disease, and pulmonary capillary hemangiomatosis.
* Persistent pulmonary hypertension of the newborn.
* Pulmonary Hypertension belonging to groups 2 to 5 of the Venice classification.
* Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C.
* Estimated creatinine clearance < 30 mL/min
* Serum aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 1.5 times the upper limit of normal.
* Hemoglobin < 75% of the lower limit of the normal range.
* Systolic blood pressure < 100 mmHg.
* Acute or chronic physical impairment (other than dyspnea), limiting the ability to comply with study requirements.
* Pregnant or breast-feeding.
* Known concomitant life-threatening disease with a life expectancy < 12 months.
* Body weight < 40 kg.
* Any condition that prevents compliance with the protocol or adherence to therapy.
* Treatment with endothelin receptor antagonists (ERAs) within 3 months prior to randomization.
* Systemic treatment within 4 week prior to randomization with cyclosporine A or tacrolimus, everolimus, sirolimus (calcineurin or mammalian target of rapamycin (mTOR) inhibitors).
* Treatment with cytochrome P3A (CYP3A) inducers within 4 weeks prior to randomization
* Known hypersensitivity to drugs of the same class as the study drug, or any of their excipients.
* Planned treatment, or treatment, with another investigational drug within 1 month prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-03 (Actual)

PRIMARY OUTCOMES:
Change in exercise pulmonary vascular resistance (PVR) | Baseline to 6 months

SECONDARY OUTCOMES:
Change in right ventricular pulmonary vascular hemodynamic coupling (RVPA). | Baseline to 6 months
Change in maximal oxygen consumption (V02 max). | Baseline to 6 months
Change in pulmonary impedance. | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Franz P. Rischard, DO, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States